CLINICAL TRIAL: NCT04050306
Title: DIMOH: New Digital Methods for Monitoring Oral Health. An in Vivo Assessment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Copenhagen (Other)
Collaborators: Innovation Fund Denmark (Individual); National and Kapodistrian University of Athens (Other); 3Shape A/S (Industry)
Responsible Party: Principal Investigator, Stavroula Michou, PhD Student, Principal Investigator, University of Copenhagen
Other Study IDs: 8053-00005B
Record Dates: First submitted 2019-08-05; First posted 2019-08-08 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Dental Caries; Tooth Wear
Keywords: Quantitative Light-Induced Fluorescence; Oral Health; Dental Caries; Tooth Wear; Optical Imaging
MeSH Terms: conditions — Dental Caries; Tooth Wear

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adolescents and young adults: Participants 12-19 years old without chronic diseases.

SUMMARY:
The objectives of this study are i) to monitor the oral health of young people over a period of one year and ii) to assess the ability of a new intraoral scanner combining fluorescence with 3D imaging to detect and monitor changes in the dental hard tissues in vivo.

The working hypotheses of this study are that i) the monitoring of oral health will benefit from using a new intraoral scanner combining fluorescence with 3D imaging and ii) the new intraoral scanner combining fluorescence with 3D imaging will aid dentists to identify changes in the dental hard tissues at earlier stages than the traditional diagnostic methods (i.e. visual-tactile, radiographic methods).

DETAILED DESCRIPTION:
Currently, monitoring oral health relies mainly on the visual examination of the oral tissues aided electively by radiographic or photographic images. In the context of oral health, monitoring involves detecting changes, sometimes rather subtle, in the soft or hard oral tissues.

The slow rate of change involved in some situations, like loss of mineral tissues due to caries or tooth wear, makes it extremely difficult for the human eye alone to identify them. It is even more challenging to accurately register and recall the original situation on the patient's follow-up visits. Clinical photographs are therefore used to aid the monitoring however, it is difficult to obtain comparable photographs from different points in time and the subjectivity involved in the process cannot be avoided.

Different criteria are used in clinical practice to register and monitor changes in the oral tissues, according to the specific condition under investigation. While identifying significant changes is an easy task, the challenge lies particularly in identifying early, incremental changes. Regarding the detection of caries lesions, a number of initial lesions typically remain unnoticed when visual examination alone is used; or even when radiographs are employed, as the latter are not sensitive to early demineralization in enamel. Concerning tooth wear (i.e. erosion, abrasion, attrition), as the gradual mineral loss occurs progressively and irreversibly, it is usually only noticed when a significant amount of hard dental tissue is already lost.

A promising clinical solution to overcome the challenges involved in the detection of early changes and monitoring of oral tissues is the use of 3D intraoral scans. Obtaining 3D scans directly from the patients (in vivo) using intraoral scanners and by comparing 3D scans obtained from the same patients at different points in time, a less subjective and more reliable comparison of data is expected: the 3D scans can be overlapped and analyzed using specific software. Therefore, it is hypothesized that 3D intraoral scans can be used for more consistent monitoring of oral health in relation to clinical photographs or clinical records.

The current 3D intraoral scanners capture the color of the oral tissues by emitting visible white light. A recently developed 3D intraoral scanner manufactured by 3Shape A/S, Denmark, is also able to emit visible blue light (415 nm wavelength) that allows capturing fluorescence from the oral tissues. Fluorescence is one of the most promising technologies for accurate detection of the early stages of enamel demineralization, but is currently available only in 1D or 2D devices. The main limitation of the existing devices featuring fluorescence, as already mentioned, is the challenge in comparing single images obtained at different points in time, which is at large influenced by imaging artifacts and noise. Imprecision in the comparison of these images compromises the ability to accurately monitor progressive demineralization of the dental hard tissues. There is no intraoral scanner reported in the scientific literature that combines fluorescence with 3D imaging. Thus, the investigators hypothesize that this new intraoral scanner will benefit the monitoring of dental hard tissues and will aid dentists to identify early changes in tissue mineralization. With this method it is only possible to examine the tooth surfaces that are visible and directly exposed into the mouth (i.e. the smooth free surfaces and the occlusal fissures); the areas between the teeth (i.e. the approximal surfaces) cannot be visualized and therefore cannot be examined using the scanner.

A total number of 70 participants will be recruited for the study, including adolescents and young adults (12-19 years old). The oral health of all participants will be examined using visual-tactile and radiographic methods. Subsequently, both the upper and lower jaw of the participants will be scanned using the intraoral scanner (TRIOS 4, 3Shape TRIOS A/S, Denmark). All participants will be monitored for 1 year with follow-up intervals of 3 to 12 months according to the risk group that they are classified into (low, moderate, high). The same clinical procedures will be followed on the follow-up examinations (3 or 6 months) as well as on the final examination (1-year follow-up) The clinical registrations from oral examination using the state-of-the-art methods (visual-tactile, radiographic) will be compared with the outcomes from the assessment using the intraoral scanner.

ELIGIBILITY:
Inclusion Criteria:

* Participants 12-19 years old without chronic diseases

Exclusion Criteria:

* Participants in need of complex dental treatment (e.g. extensive restorative work, extractions, prosthetic treatment).
* Participants using partial/complete removable dentures or other appliances (i.e. orthodontic).

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The participants in this project will be healthy young people 12-19 years old. The adolescents (12-16 years old) will be recruited in Denmark and they will be students from national public schools in the Capital Region of Denmark.
  The young adults (18-19 years old) will be recruited in Greece and they will be 1st-year University students at the School of Dentistry of the National and Kapodistrian University of Athens.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2019-03-27 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-12-18 (Estimated)

PRIMARY OUTCOMES:
1st Clinical caries score | Baseline
  Caries score registered by conducting the traditional clinical (visual-tactile) and radiographic examination.
  The International Caries Detection and Assessment System (ICDAS) codes will be used. Scale ranges from 0 (sound surfaces) to 6 (extensive cavitated caries lesions located into the inner third of the dentin).
1st Scanner caries score | Baseline
  Caries score registered using the intraoral scanner and the accompanying software (Trios, 3Shape TRIOS A/S, Denmark) which will provide an automated caries score.
  Scale used:
  0 (sound surfaces),
  1. (initial caries lesions in enamel or into the outer third of dentin),
  2. (moderate - extensive caries lesions located into the middle - inner third of dentin).
2nd Clinical caries score | 3 or 6 months after the baseline examination dependent on the risk of the patient (i.e. 3 months for high risk, 6 months for moderate risk, NO 2nd clinical caries score for low risk)
  Caries score registered by conducting the traditional clinical (visual-tactile) and radiographic examination.
  The International Caries Detection and Assessment System (ICDAS) codes will be used.
  Scale ranges from 0 (sound surfaces) to 6 (extensive cavitated caries lesions located into the inner third of the dentin).
2nd Scanner caries score | 3 or 6 months after the baseline examination dependent on the caries risk of the patient (i.e. 3 months for high risk, 6 months for moderate risk, NO 2nd score for low risk)
  Caries score registered using the intraoral scanner and the accompanying software (Trios, 3Shape TRIOS A/S, Denmark) which will provide an automated caries score.
  Scale used:
  0 (sound surfaces),
  1. (initial caries lesions in enamel or into the outer third of dentin),
  2. (moderate - extensive caries lesions located into the middle - inner third of dentin).
3rd Clinical caries score | 12 months after the baseline examination
  Caries score registered by conducting the traditional clinical (visual-tactile) and radiographic examination.
  The International Caries Detection and Assessment System (ICDAS) codes will be used.
  Scale ranges from 0 (sound surfaces) to 6 (extensive cavitated caries lesions located into the inner third of the dentin).
3rd Scanner caries score | 12 months after the baseline examination
  Caries score registered using the intraoral scanner and the accompanying software (Trios, 3Shape TRIOS A/S, Denmark) which will provide an automated caries score.
  Scale used:
  0 (sound surfaces),
  1. (initial caries lesions in enamel or into the outer third of dentin),
  2. (moderate - extensive caries lesions located into the middle - inner third of dentin).
1st Tooth wear scan score | Baseline
  Tooth wear score is registered by visually examining the 3D scans of the participants and applying the Basic Erosive Wear Examination (BEWE) index.
  Scale ranges from 0 (No surface loss) to 3 (Distinct defect, hard tissue loss of more than 50% of the surface area).
1st Clinical tooth wear score | Baseline
  Tooth wear score is registered by examining the participants clinically and applying the Basic Erosive Wear Examination (BEWE) index.
  Scale ranges from 0 (No surface loss) to 3 (Distinct defect, hard tissue loss of more than 50% of the surface area).
2nd Tooth wear scan score | 3 or 6 months after the baseline examination dependent on the risk of the patient (i.e. 3 months for high risk, 6 months for moderate risk, NO 2nd score for low risk)
  Tooth wear score is registered by visually examining the 3D scans of the participants and applying the Basic Erosive Wear Examination (BEWE) index.
  Scale ranges from 0 (No surface loss) to 3 (Distinct defect, hard tissue loss of more than 50% of the surface area).
2nd Clinical tooth wear score | 3 or 6 months after the baseline examination dependent on the risk of the patient (i.e. 3 months for high risk, 6 months for moderate risk, NO 2nd score for low risk)
  Tooth wear score is registered by examining the participants clinically and applying the Basic Erosive Wear Examination (BEWE) index.
  Scale ranges from 0 (No surface loss) to 3 (Distinct defect, hard tissue loss of more than 50% of the surface area).
3rd Tooth wear scan score | 12 months after the baseline examination
  Tooth wear score is registered by visually examining the 3D scans of the participants and applying the Basic Erosive Wear Examination (BEWE) index.
  Scale ranges from 0 (No surface loss) to 3 (Distinct defect, hard tissue loss of more than 50% of the surface area).
3rd clinical tooth wear score | 12 months after the baseline examination
  Tooth wear score is registered by examining the participants clinically and applying the Basic Erosive Wear Examination (BEWE) index.
  Scale ranges from 0 (No surface loss) to 3 (Distinct defect, hard tissue loss of more than 50% of the surface area).
Tooth surface change due to tooth wear at 12 months | Baseline - 12 months
  The 3D models of the same participants at two different points in time (baseline and 12-month follow-up examination) will be supperimposed and possible tooth surface differences between the 2 models will be quantified using specific software (Trios Patient Monitoring, 3Shape TRIOS A/S, Denmark).
  The maximum difference value per tooth will be registered in mm (measurement error 0.05 mm).

CONTACTS AND LOCATIONS:
Overall Officials: STAVROULA MICHOU, DDS, Principal Investigator — Department of Odontology, University of Copenhagen
Locations (2):
- Department of Odontology, Faculty of Health and Medical Sciences, Univeristy of Copenhagen, Copenhagen, Denmark
- School of Dentistry, National and Kapodistrian Univeristy of Athens, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pitts NB, Zero DT, Marsh PD, Ekstrand K, Weintraub JA, Ramos-Gomez F, Tagami J, Twetman S, Tsakos G, Ismail A. Dental caries. Nat Rev Dis Primers. 2017 May 25;3:17030. doi: 10.1038/nrdp.2017.30. PMID 28540937
- [Background] Ganss C, Lussi A. Diagnosis of erosive tooth wear. Monogr Oral Sci. 2014;25:22-31. doi: 10.1159/000359935. Epub 2014 Jun 26. PMID 24993255
- [Background] Marro F, De Lat L, Martens L, Jacquet W, Bottenberg P. Monitoring the progression of erosive tooth wear (ETW) using BEWE index in casts and their 3D images: A retrospective longitudinal study. J Dent. 2018 Jun;73:70-75. doi: 10.1016/j.jdent.2018.04.008. Epub 2018 Apr 13. PMID 29660487
- [Background] Pretty IA. Caries detection and diagnosis: novel technologies. J Dent. 2006 Nov;34(10):727-39. doi: 10.1016/j.jdent.2006.06.001. Epub 2006 Aug 9. PMID 16901606
- [Background] Pretty IA, Ellwood RP. The caries continuum: opportunities to detect, treat and monitor the re-mineralization of early caries lesions. J Dent. 2013 Aug;41 Suppl 2:S12-21. doi: 10.1016/j.jdent.2010.04.003. PMID 23985434
- [Background] Gomez J, Zakian C, Salsone S, Pinto SC, Taylor A, Pretty IA, Ellwood R. In vitro performance of different methods in detecting occlusal caries lesions. J Dent. 2013 Feb;41(2):180-6. doi: 10.1016/j.jdent.2012.11.003. Epub 2012 Nov 9. PMID 23146817
- [Background] Pitts NB, Ekstrand KR; ICDAS Foundation. International Caries Detection and Assessment System (ICDAS) and its International Caries Classification and Management System (ICCMS) - methods for staging of the caries process and enabling dentists to manage caries. Community Dent Oral Epidemiol. 2013 Feb;41(1):e41-52. doi: 10.1111/cdoe.12025. PMID 24916677
- [Background] Bartlett D, Ganss C, Lussi A. Basic Erosive Wear Examination (BEWE): a new scoring system for scientific and clinical needs. Clin Oral Investig. 2008 Mar;12 Suppl 1(Suppl 1):S65-8. doi: 10.1007/s00784-007-0181-5. Epub 2008 Jan 29. PMID 18228057
- [Background] Norrisgaard PE, Qvist V, Ekstrand K. Prevalence, risk surfaces and inter-municipality variations in caries experience in Danish children and adolescents in 2012. Acta Odontol Scand. 2016;74(4):291-7. doi: 10.3109/00016357.2015.1119306. Epub 2015 Dec 14. PMID 26651538
- [Derived] Michou S, Tsakanikou A, Bakhshandeh A, Ekstrand KR, Rahiotis C, Benetti AR. Occlusal caries detection and monitoring using a 3D intraoral scanner system. An in vivo assessment. J Dent. 2024 Apr;143:104900. doi: 10.1016/j.jdent.2024.104900. Epub 2024 Feb 25. PMID 38412900

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-08): https://cdn.clinicaltrials.gov/large-docs/06/NCT04050306/Prot_SAP_000.pdf